CLINICAL TRIAL: NCT06388954
Title: Effect of Trans-auricular Vagus Nerve Stimulation on Plasticity Biomarkers,Interleukin-6 and Motor Performance Post Stroke : A Randomized Controlled Clinical Trial
Brief Title: Plasticity Biomarkers,Interleukin-6 and Motor Performance in Response to Vagus Nerve Stimulation After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005107
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Motor Disorders
Keywords: Neurotrophic Factors; Ischemic Stroke; Neural Plasticity; Interleukin-6; Vagus Nerve Stimulation
MeSH Terms: conditions — Stroke; Motor Disorders; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized controlled study.
Who Masked: Participant
Masking Description: Patients participated will be masked about the type of intervention, where (GA) patients will receive physical therapy program + sham transcutaneous auricular Vagus nerve stimulation, while patients in (GB) will receive true transcutaneous auricular Vagus nerve stimulation in addition to the same physical therapy program as (GA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (GA) (Placebo Comparator): Patients in the control group (GA) will be treated by 12 sessions of sham transcutaneous auricular Vagus nerve stimulation for 30 minutes immediately, will be followed by 30 minutes of a selected physical therapy program, three sessions per week for four consecutive weeks. Sham transcutaneous vagal nerve stimulation was performed using the same procedures as the study group but without electrical stimulation.
  Interventions: Device: Sham Trancutaneous auricular Vagus Nerve Stimulation
- Study group (GB) (Experimental): Patients in the study group (GB) will be treated by 12 sessions of true transcutaneous auricular Vagus nerve stimulation for 30 minutes , then immediately followed by 30 minutes of a selected physical therapy program (GA), three sessions per week for four consecutive weeks. The stimulation of the auricular branch of the Vagus nerve will be performed by conventional TENS device with one channel and two electrodes.
  Interventions: Device: True Transcutaneous auricular Vagus Nerve Stimulation (TaVNS)

INTERVENTIONS:
Device: True Transcutaneous auricular Vagus Nerve Stimulation (TaVNS) — Vagus Nerve Stimulation (VNS) consists in the activation of the Vagus nerve using electrical current, Transcutaneous auricular VNS works through the placement of noninvasive electrodes on the neck or auricle for stimulation of the auricular branch of the vagus nerve.
  Transcutaneous electrical nerve stimulation (TENS) electrodes will be used to stimulate the auricular branch of the Vagus nerve, The active electrode will be placed on the cymba concha of the left ear. This reduced the risk of taVNS side eﬀect on the heart. The reference electrode will be placed outside the left ear attached to the tragus. TENS parameters used were: 30 minutes treatment time, a pulse width of 300 microseconds, pulse frequency 20 hertz and a duty cycle of 25%. The stimulation intensity was set at super-threshold levels, such as 200% of patient perceptual threshold.
  Other Names: Transcutaneous Vagus Nerve Stimulation (TVNS)
  Arms: Study group (GB)
Device: Sham Trancutaneous auricular Vagus Nerve Stimulation — Sham transcutaneous vagal nerve stimulation will be performed by the same procedures of the study group but without electrical stimulation. The active electrodes will be attached to the left cymba conchae. The taVNS stimulator will be turned on and the stimulation intensity will be increased until the patient perceived the electrical stimulation and then the stimulator will be turned off.
  Arms: Control group (GA)

SUMMARY:
Seventy-eight clinically verified Egyptian patients from both sexes with ischemic stroke that occurred at least 6 months to 2 years before inclusion will be randomly assigned into 2 groups, control group (GA) and the experimental group (GB). Patients will be randomly assigned into two equal groups: the control group (GA) and the experimental group (GB). Patients in the control group (GA) will be treated with sham Vagus nerve stimulation (taVNS) immediately before a selected physical therapy program, while in the experimental group (GB), patients will receive real transcutaneous auricular Vagus nerve stimulation (taVNS) followed by the same selected physical therapy program as (GA). Plasma level of Brain-Derived Neurotrophic Factors (BDNF) and Interleukin-6 (IL-6), Box and Blocks Test (BBT), and modified Ashworth scale (MAS) will be assessed at baseline and immediately post-treatment.

DETAILED DESCRIPTION:
Background: Neuromodulation techniques play an integral role in restoring motor function in stroke patients by affecting the adaptive neuroplasticity and activation of neuromodulators that may reduce brain inflammation post stroke.

Objective: To assess the efficacy of transcutaneous auricular vagal nerve stimulation on plasma levels of Brain-Derived Neurotrophic Factors (BDNF), Interleukin-6 (IL-6), gross manual dexterity, and muscle tone in patients with ischemic stroke.

Materials and Methods: Seventy-eight clinically verified Egyptian patients from both sexes with ischemic stroke that occurred at least 6 months to 2 years before inclusion, aged 55 to 65 years, were recruited. Patients will be randomly assigned into two equal groups; control group (GA) and the experimental group (GB). Patients in the control group (GA) were treated with sham Vagus nerve stimulation (taVNS) immediately before a selected physical therapy program, while in the experimental group (GB), patients received real transcutaneous auricular Vagus nerve stimulation (taVNS) followed by the same selected physical therapy program as (GA). Plasma levels of Brain-Derived Neurotrophic Factors (BDNF), serum Interleukin-6 (IL-6) , Box and Blocks Test (BBT) and Modified Ashworth scale (MAS) were assessed at baseline and immediately post-treatment.

Results: There was a statistically significant improvement in BBT, plasma IL-18 level and BDNF in experimental group (GB) post-treatment (P< 0.05) with no change in MAS. There was no statistical significant difference in BBT, plasma Interleukin-6 (IL-6) and MAS in control group post treatment (P> 0.05). While, there is a statistically significant improvement in BDNF in the control group post treatment. A statistically significant improvement was observed of BBT and BDNF in the study group compared to the control group (P< 0.05). There was no statistical significant difference in MAS between study and control groups (P> 0.05).

Conclusions: Non-invasive VNS as an adjunct to conventional physical rehabilitation enhances neuroplasticity and improves upper limb motor ability after ischemic stroke, as well as reducing the stroke-induced inflammatory process, which may affect the disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic patients with ischemic middle cerebral artery stroke
* The duration of illness ranged from at least 6 months to 2 years after stroke.
* Patient's age ranged from 55 to 65 years, patients with unilateral upper limb motor function impairment.
* Patients able to transfer at least one block in Box and Blocks Test.
* Patients with sufficient cognitive abilities that enables them to understand and follow instructions.
* Spasticity of upper limb muscles ranged from (grade 1:2) according to Modified Ashworth scale.

Exclusion Criteria:

* Other neurological diseases that affect upper limb function other than stroke (e.g.: Multiple sclerosis, peripheral neuropathy, Parkinsonism….etc.).
* Hemorrhagic stroke
* Visual or auditory impairment affecting their ability to complete the testing.
* Cognitive impairment.
* Cardiovascular problems and pulmonary or kidney disorders
* Musculoskeletal disorders (e.g. scoliosis, kyphosis, severe arthritis…etc.)
* Severe spasticity (a Modiﬁed Ashworth Scale score ≥3).
* Patients with any taVNS contraindications such as previous surgical intervention on Vagus nerve.
* Low blood pressure (<100/60mmHg) or low heart rate (<60bpm) and or high blood pressure (>220/130 mmHg).
* Pacemaker or other implanted electrical device.
* Any current or past history of cardiovascular disorders
* Facial or ear pain
* Recent ear trauma .

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Muscle tone of the upper limb | Baseline Assessment and Immediately Post Treatment.
  The Modified Ashworth Scale (MAS) will be used; it is a six-point ordinal scale. It ranges from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). The muscle tone was measured by observing the response of the muscle group to the resistance of passive movement in the affected hand. The degree of muscle tone in the affected hand was classified as (0 = normal, 1 or 1+ = mild, 2 or 3 = moderate, or 4 = severe).
Gross hand dexterity | Baseline Assessment and Immediately Post Treatment.
  The Box and Blocks Test (BBT) will be used; it is a quick, simple, and inexpensive test for measuring unilateral gross manual dexterity in stroke. The patients were asked to transfer as many blocks as they could from one compartment to the other for 60 seconds. The patient was allowed to choose any block of any color and to carry only one block each time with his hand, which must cross over the partition.
Level of Plasma brain-derived Derived factor (BDNF) | Baseline Assessment and Immediately Post Treatment.
  Sandwich-ELISA kits will be used according to the manufacturer's instructions. Venous blood samples were collected in a disposable plastic vacuum tube with an anticoagulant. Samples were centrifuged for 15 min at 1000×g at 2-8 °C within 30 min of collection.
Level of Serum Interleukin IL-6 | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  Interleukin-6 (IL-6) is a crucial inflammatory factor in that its significant increase was observed in stroke patients shortly following the ischemic event and serves a vital role as a messenger molecule between leucocytes, the vascular endothelium, and parenchyma. A single referral lab will test the samples using ELISA and U/CyTech kits. From each participant, 10 milliliters of non-fasting blood sample will be obtained 6 to 24 hours after the onset of symptoms and kept in citrate tubes. Blood samples will thereafter centrifuged within 1 hour at 3000 × g for 15 minutes at 4°C and resultant plasma will be kept in -80°C.

CONTACTS AND LOCATIONS:
Overall Officials: Engy B Saleh, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No